CLINICAL TRIAL: NCT01282229
Title: A Multi-Center Single Blind Study of the Laser Assisted New Attachment Procedure Compared to Scaling and Root Planing Alone, Modified Widman Flap Surgery, and Coronal Debridement Alone in the Treatment of Chronic Periodontitis
Brief Title: Study to Compare Laser Assisted New Attachment Procedure (LANAP) to Traditional Treatments of Chronic Periodontitis
Acronym: LANAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute for Advanced Laser Dentistry (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MDT MC 06-001
Record Dates: First submitted 2011-01-13; First posted 2011-01-24 (Estimated); Results first posted 2015-10-14 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Periodontitis
Keywords: LANAP, Laser dentistry
MeSH Terms: conditions — Chronic Periodontitis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- LANAP Quadrant (Active Comparator): Treated with LANAP
  Interventions: Device: LANAP
- Modified Widman Flap (No Intervention): Quadrant treated with Modified Widman Flap surgery
- Scaling and Root Planing (No Intervention): Quadrant treated with scaling and root planing alone
- Coronal Debridement (No Intervention): Quadrant treated with coronal debridement

INTERVENTIONS:
Device: LANAP — Laser Assisted New Attachment Procedure (LANAP protocol) using the FR Pulsed Nd:YAG laser
  Other Names: Periolase MVP 7
  Arms: LANAP Quadrant

SUMMARY:
The purpose of this study is to compare the Laser Assisted New Attachment Procedure (LANAP protocol) using the Free-running (FR) Pulsed Neodimium: Yttrium aluminium garnet (Nd:YAG) laser to Scaling and Root Planing (SRP) alone, Modified Widman Flap (MFF) surgery, and Coronal Debridement (CD) alone with respect to periodontal clinical attachment level gain.

DETAILED DESCRIPTION:
This multi-center study of the Laser Assisted New Attachment Procedure (LANAP protocol) using the FR Pulsed Nd:YAG laser compared to Scaling and Root Planing alone, Modified Widman Flap (MWF) surgery, and Coronal Debridement (CD) alone will utilize a single-blind, four-quadrant split-mouth design with MWF as the positive control, CD as a weak positive control and SRP as the standard treatment control. The study will be conducted at three (3) to five (5) investigational centers. Subjects will receive the Laser Assisted New Attachment Procedure (LANAP protocol) using the pulsed FR Nd:YAG laser, Scaling and Root Planing alone, Modified Widman Flap surgery, and Coronal Debridement alone each in one quadrant of their mouth at Baseline. Treatment modalities are randomly assigned to quadrants at the time of treatment.

Efficacy evaluations, including clinical attachment level (CAL), probing depth (PD), and bleeding on probing (BOP) will be performed at Baseline, month 6, and month 12 using a Florida Electronic Probe. Radiographs will be taken at Screening/Baseline and at month 6 and month 12.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects will have chronic adult periodontitis as characterized by all four quadrants of the mouth.
2. Subjects will be 25-75 years of age.
3. Subjects will be able to follow verbal and/or written instructions, perform Oral Hygiene according to the protocol, and return to the center for specified study visits.
4. Subjects must have had no subgingival scaling instrumentation including scaling and root planing, regular periodontal maintenance procedures or any subgingival cleaning < 12 (twelve) months prior to Baseline examination.
5. Subjects must have had no history of periodontal surgical procedures of any type prior to Baseline examination.
6. Subjects must be non-smokers of any type or former smokers (>6 (six) months stopped), and not using or taking any nicotine product.
7. Subjects will have clinical and/or radiographic evidence of subgingival calculus in each quadrant.
8. Subjects have no more than one missing tooth per quadrant, excluding 3rd molars.
9. Subjects will be able to sign the informed consent form.

Exclusion Criteria:

1. Subject receiving subgingival scaling instrumentation including scaling and root planing, regular periodontal maintenance procedures or any subgingival cleaning less than twelve (12) months prior to Baseline examination.
2. Subjects receiving periodontal surgery of any type prior to Baseline examination.
3. Subjects with dental implants.
4. Subjects with a compromised heart condition, history of rheumatic fever, or joint replacement requiring prophylaxis.
5. Subjects having taken systemic cancer therapy and/or radiation therapy at any time
6. Subjects with clinically significant acute or concurrent illness
7. Subjects with clinically significant chronic illness.
8. Subjects with a disease of the connective tissue.
9. Subjects taking medications which are likely to cause gingival hyperplasia, within ONE MONTH prior to Baseline examination
10. Subjects taking antimicrobials within ONE MONTH prior to Baseline examination
11. Subjects taking non-steroidal anti-inflammatory drugs at a therapeutic dose within the TWO WEEKS prior to Baseline examination.
12. Subjects taking steroids of any kind within ONE MONTH prior to baseline examination.
13. Subjects taking continuous low doses of tetracycline within THREE MONTHS prior to Baseline examination
14. Subjects taking an investigational drug within TWO MONTHS prior to Baseline examination
15. Subjects taking or having taken bisphosphonates of any kind for any reason.
16. Female, nonsterile subjects who are pregnant or lactating.
17. Subjects who, in the investigator's opinion, would not comply with the study procedures.
18. Smokers of any type or former smokers and subjects that take or use any nicotine product.
19. Excessive alcohol intake.
20. No current restorative or endodontic treatment needs

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Actual)
Dates: Start 2010-10; Primary Completion 2014-03 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymund A Yukna, DMD, MS, Study Director — University of Colorado Scholl of Dentistry; Henry Greenwell, DMD. MSD, Principal Investigator — University of Louisville, School of Dentistry; Mark Reynolds, DDS, PhD, Principal Investigator — University of Maryland, School of Dentistry; James Finley, DMD, Principal Investigator — Finley Periodontics; Thomas McCawley, DDS, Principal Investigator — McCawly & DeTure
Locations (1):
- University of Colorado, Denver, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- All Participants: Subjects will receive the Laser Assisted New Attachment Procedure (LANAP protocol) using the pulsed FR Nd:YAG laser, Scaling and Root Planing alone, Modified Widman Flap surgery, and Coronal Debridement alone each in one randomized quadrant of their mouth at Baseline.
Period: Overall Study
Arm/Group | All Participants
Started | 59 (59 Participants contributed 236 quadrants (59*4))
Completed | 57 (57 Participants contributed 228 quadrants (57*4))
Not Completed | 2
Not completed — Protocol Violation | 2

BASELINE CHARACTERISTICS:
Population: Data are for number of quadrants
Arm/Group | All Participants
Number analyzed (Participants) | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 51
  >=65 years | 6
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27
  Male | 30
Average Probing Depth (PD) [Mean (Standard Deviation); unit: mm]
  PD = 5-6mm (LANAP Quadrant) | 5.364 (.553)
  PD = 5-6mm ( Modified Widman Flap) | 5.358 (.569)
  PD = 5-6mm (Scaling and Root Planing) | 5.358 (.570)
  PD = 5-6mm (Coronal Debridement) | 5.382 (.554)
  PD >= 7mm (LANAP Quadrant) | 7.606 (.867)
  PD >= 7mm (Modified Widman Flap) | 7.562 (.901)
  PD >= 7mm (Scaling and Root Planing) | 7.657 (.967)
  PD >= 7mm (Coronal Debridement) | 7.672 (1.069)
Average Clinical Attachment Level (CAL) [Mean (Standard Deviation); unit: mm]
  PD = 5-6mm (LANAP Quadrant) | 5.431 (1.301)
  PD = 5-6mm ( Modified Widman Flap) | 5.440 (1.349)
  PD = 5-6mm (Scaling and Root Planing) | 5.364 (1.244)
  PD = 5-6mm (Coronal Debridement) | 5.468 (1.486)
  PD >= 7mm (LANAP Quadrant) | 7.453 (1.594)
  PD >= 7mm (Modified Widman Flap) | 7.737 (1.586)
  PD >= 7mm (Scaling and Root Planing) | 7.528 (1.751)
  PD >= 7mm (Coronal Debridement) | 7.681 (1.659)
Bleeding on Probing (BOP) [Mean (Standard Deviation); unit: percentage of pockets] — Percent of pockets within a quadrant that bled on probing by time and treatment
  percentage of pockets
    LANAP Quadrant | 49.4 (31.4)
    Modified Widman Flap | 46.5 (31.2)
    Scaling and Root Planing | 48.2 (30.6)
    Coronal Debridement | 47.5 (31.2)
Gingival Index (GI) [Mean (Standard Deviation); unit: units on a scale] — Modified Gingival Index of Lobene et al (1986). Inflammation rated 0 (none) to 4 (severe).
  units on a scale
    LANAP Quadrant | 2.48 (0.95)
    Modified Widman Flap | 2.42 (0.95)
    Scaling and Root Planing | 2.44 (0.96)
    Coronal Debridement | 2.43 (0.95)

OUTCOME MEASURES:

1. Primary Outcome: Gain in Clinical Attachment Level of Periodontal Tissues
Description: Periodontitis causes loss of attachment of the tooth root to the surrounding bone. Change in Clinical Attachment Level (CAL) estimates the number of mm's of reattachment gained as a result of the treatment.
Time Frame: Baseline, 6, 12 months
Population: 5-6 mm baseline PD partition had a different sample size than the 7+mm partition.
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: pockets
Groups:
- LANAP Quadrant (5-6mm Pockets); LANAP Quadrant (≥7mm Pockets): Treated with LANAP
  LANAP: Laser Assisted New Attachment Procedure (LANAP protocol) using the FR Pulsed Nd:YAG laser
- Modified Widman Flap (5-6mm Pockets); Modified Widman Flap (≥7mm Pockets): Quadrant treated with Modified Widman Flap surgery
- Scaling and Root Planing (5-6mm Pockets); Scaling and Root Planing (≥7mm Pockets): Quadrant treated with scaling and root planing alone
- Coronal Debridement (5-6mm Pockets); Coronal Debridement (≥7mm Pockets): Quadrant treated with coronal debridement
Arm/Group | LANAP Quadrant (5-6mm Pockets) | LANAP Quadrant (≥7mm Pockets) | Modified Widman Flap (5-6mm Pockets) | Modified Widman Flap (≥7mm Pockets) | Scaling and Root Planing (5-6mm Pockets) | Scaling and Root Planing (≥7mm Pockets) | Coronal Debridement (5-6mm Pockets) | Coronal Debridement (≥7mm Pockets)
Number analyzed (Participants) | 52 | 51 | 52 | 51 | 52 | 51 | 52 | 51
Number analyzed (pockets) | 445 | 234 | 434 | 224 | 495 | 239 | 439 | 210
mm
  Change in CAL @ 6 mo | 1.361 (1.736) | 2.387 (2.038) | 1.180 (1.587) | 2.329 (1.909) | 1.347 (1.833) | 2.061 (2.243) | 0.796 (1.723) | 1.573 (1.945)
  Change in CAL @ 12 mo | 1.498 (1.638) | 2.458 (2.005) | 1.229 (1.588) | 2.120 (1.840) | 1.425 (1.810) | 2.330 (2.137) | 1.033 (1.857) | 1.762 (2.082)

2. Secondary Outcome: Change in Probing Depth (PD)
Description: Positive numbers indicate average decrease in probing depth (improvement).
Time Frame: Baseline, 6, 12 months
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: pockets
Arm/Group | LANAP Quadrant | Modified Widman Flap | Scaling and Root Planing | Coronal Debridement
Number analyzed (Participants) | 57 | 57 | 57 | 57
Number analyzed (pockets) | 487 | 459 | 527 | 476
mm
  5-6mm @ 6 mo | 1.674 (1.402) | 1.834 (1.263) | 1.550 (1.486) | 1.084 (1.544)
  5-6mm @ 12 mo | 1.888 (1.446) | 1.831 (1.305) | 1.702 (1.556) | 1.223 (1.749)
  >=7mm @ 6 mo | 2.716 (1.832) | 3.117 (1.585) | 2.525 (1.897) | 1.976 (1.773)
  >=7mm @ 12 mo | 3.097 (1.766) | 3.004 (1.581) | 2.846 (2.001) | 2.108 (1.959)

3. Secondary Outcome: Change in Bleeding on Probing (BOP)
Description: Percent of pockets within a quadrant that changed from baseline to 6 or 12 months. Negative numbers are a decrease in bleeding on probing which represents clinical improvement.
  Each quadrant within the patient represents one of four treatments, the unit of analysis. Pockets are replications within treatments and vary in number among quadrants.
Time Frame: Baseline, 6, 12 months
Measure: Mean (Standard Deviation); unit: percentage of pockets that bled
Units Other Than Participants: quadrants
Arm/Group | LANAP Quadrant | Modified Widman Flap | Scaling and Root Planing | Coronal Debridement
Number analyzed (Participants) | 57 | 57 | 57 | 57
Number analyzed (quadrants) | 57 | 57 | 57 | 57
percentage of pockets that bled
  change @ 6 mo | -24.9 (32.7) | -22.9 (30.7) | -23.7 (28.0) | -18.0 (31.2)
  change @ 12mo | -23.0 (29.7) | -20.4 (28.2) | -20.1 (27.7) | -15.7 (28.4)

4. Secondary Outcome: Change in Gingival Index
Description: The gingival index is a 0-4 unit scale that the examiner uses to estimate the amount of edema and erythema at 2 locations (lingual and buccal) for every tooth in the quadrant. Zero (0) represents no redness and swelling and four (4) represents severe redness and swelling. Negative numbers are a decrease in in examiner estimate of erythema and edema and represent an improvement in clinical outcome.
Time Frame: Baseline, 6, 12 months
Measure: Mean (Standard Deviation); unit: units on a scale from 0-4
Units Other Than Participants: locations
Arm/Group | LANAP Quadrant | Modified Widman Flap | Scaling and Root Planing | Coronal Debridement
Number analyzed (Participants) | 57 | 57 | 57 | 57
Number analyzed (locations) | 832 | 819 | 823 | 810
units on a scale from 0-4
  6 months | -1.28 (1.28) | -1.30 (1.31) | -1.28 (1.27) | -1.14 (1.28)
  12 months | -1.29 (1.19) | -1.27 (1.22) | -1.26 (1.20) | -1.14 (1.22)

5. Secondary Outcome: Discomfort
Description: Subjects recorded in a diary discomfort on a 10 point visual analog scale daily for the week following treatment. Subjects provided an estimate for each of the four treated quadrants. Zero (0) represents no pain or discomfort and ten (10) represents severe pain and/or discomfort. For each subject discomfort scores on each day from Day 1 to Day 7 were summed. Medians and ranges for each treatment are recorded. The total score could range from 0 to 70.
Time Frame: 1-7 days
Population: Subjects with missing data (e.g., missing diary entries) are not included in the analysis.
Measure: Median (Full Range); unit: sum of units on a scale
Units Other Than Participants: quadrants
Arm/Group | LANAP Quadrant | Modified Widman Flap | Scaling and Root Planing | Coronal Debridement
Number analyzed (Participants) | 54 | 53 | 54 | 53
Number analyzed (quadrants) | 54 | 53 | 54 | 53
sum of units on a scale | 10 [0 to 60.5] | 19 [0 to 56] | 4.4 [0 to 61.5] | 3.5 [0 to 68.5]

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | LANAP Quadrant | Modified Widman Flap | Scaling and Root Planing | Coronal Debridement
Serious Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59
Other Adverse Events (participants affected / at risk) | 0/59 | 0/59 | 0/59 | 0/59

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No